CLINICAL TRIAL: NCT03892265
Title: A Longitudinal Cohort Study to Evaluate Cardiovascular Risk Factors and Disease in Haiti
Status: Active, not recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1803019037; R01HL143788 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypertension; Diabetes; Obesity; Kidney Diseases; Dyslipidemias; Smoking; Alcohol Use, Unspecified; Physical Inactivity; Poor Diet; Inflammation; Myocardial Infarction; Heart Failure; Stroke; Cardiac Death
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Obesity; Kidney Diseases; Dyslipidemias; Smoking; Alcohol Drinking; Sedentary Behavior; Inflammation; Myocardial Infarction; Heart Failure; Stroke; Death | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biologic specimens include blood and urine specimens. A blood sample will be assessed for hematology, serum creatinine, glucose, cholesterol, and lipids (high-density lipoprotein and low-density lipoprotein), HIV-1, and finger prick lead level at the GHESKIO laboratory at baseline. Serum creatinine, glucose, cholesterol and lipids will be repeated at 24 months, and thereafter every 2 years. A urine sample will be assessed for a urine albumin to creatinine ratio (ACR) using urine supernatant samples at enrollment and 24 months, and every 2 years thereafter. Biobanked specimens (whole blood, plasma, urine, stool) will be collected on all participants at enrollment and at 24 months (blood only). At 48 and 72 months fasting blood and urine will be biobanked, along with stool at 72 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Study — No intervention is included in this observational study.

SUMMARY:
Investigators will establish a longitudinal cohort of ~3,000 adults >18 years in Port-au-Prince using multistage random sampling, and follow them longitudinally to evaluate the prevalence and incidence of cardiovascular disease risk factors and diseases. Cardiovascular risk factors include hypertension, diabetes, obesity, dyslipidemia, kidney disease, poor diet, cigarette smoking, physical inactivity, and inflammation. Cardiovascular disease include angina and myocardial infarction, heart failure, stroke, and CVD mortality. It is anticipated that hypertension prevalence will be ≥10% in 18-30 year olds, that hypertension incidence will be >10 events/1000 person years. Association of determinants and risk factors with CVD will also be examined. Whole blood, serum, plasma, stool, and urine samples will be biobanked for future studies.

DETAILED DESCRIPTION:
Investigators propose a longitudinal observational study which includes establishing a population-based longitudinal cohort to determine the prevalence and incidence of cardiovascular risk factors and diseases in Haiti. Cardiovascular risk factors include hypertension, diabetes, obesity, kidney disease, dyslipidemia, smoking, alcohol use, physical inactivity, poor diet, and inflammation. Cardiovascular diseases include angina and myocardial infarction, heart failure, stroke and cardiac death. The cohort will include ~3,000 adults (>18 years) living in Port-au-Prince who will be followed longitudinally. Participants will be selected via multistage random sampling using census blocks . The GHESKIO Community Advisory Board and GHESKIO community health workers (CHWs) will conduct community sensitization about the study prior to study recruitment. CHWs will introduce the study to selected households and individuals, who will then be referred to the research team at GHESKIO for informed consent and study enrollment procedures. Participants will complete the study enrollment, 12- and 24-month, in addition to subsequent annual study visits at GHESKIO. These study visits include a study questionnaire, measurement of blood pressure and assessment for cardiovascular symptoms and events. Laboratory measures and an electrocardiogram will be done at study enrollment and the 24-month visit, and subsequently every 2 years. Participants will also provide blood, urine and stool samples for biobanking at study enrollment. Blood and urine will be collected at 24, 48 and 72 months, with stool also collected at 72 months. CHWs will perform home visits every 6 months on all participants to update locator information, measure blood pressure, and ask about cardiovascular symptoms and events. CHWs will also call the participant every three months to confirm contact information. Any participant who reports a cardiovascular symptom or event to research staff at any time during the study will be referred to the GHESKIO clinic or to a GHESKIO-affiliate hospital for clinical care. The research team will abstract data from medical records of referred patients on information regarding diagnosis codes, laboratory results, diagnostic imaging and cause of death.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 years, primary residence in the study area of Port-au-Prince (defined as having slept at the household at least once in the past two weeks and considers the household their primary residence with no plans to move in the next 24 months),
* able to provide consent for study procedures,
* agrees to study procedures, and
* willing to be contacted at a new residence if a move occurs

Exclusion Criteria:

* serious medical conditions or cognitive impairment preventing study participation as judged by research physicians,
* unable to speak and understand French or Creole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 3,000 adults >=18 years from a population-representative sample. Participants will be selected via multistage random sampling. Investigators will randomly select approximately 2,045 GPS waypoints across census blocks with the number of waypoints per block proportional to the IHSI estimated population size of each block. GPS waypoints will be randomly selected from satellite area maps, using ArcGIS software, and identified with GPS devices.
Sampling Method: Probability Sample
Enrollment: 3005 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CVD risk factors and diseases and their association with social and environmental determinants in an established longitudinal cohort of ~3,000 Haitian adults | Baseline
  The prevalence of CVD risk factors including HTN, diabetes, obesity, cigarette smoking, dyslipidemia, kidney disease, poor diet, physical inactivity, and inflammation will be calculated. Prevalence will be reported for categorical risk factors (e.g., HTN), and mean and standard deviation will be estimated for continuous risk factors (e.g., BP, lipid levels). The research team will also estimate the prevalence of each CVD outcome including MI, HF, and stroke.

SECONDARY OUTCOMES:
Incidence of CVD risk factors and CVD during ~7 years of follow-up and their association with social and environmental determinants | Participants will be followed for ~7 years
  Investigators will calculate the incidence rate of each CVD risk factor per 1000 person years (PY) of follow-up among participants without the respective CVD risk factor at baseline using a Horvitz-Thompson type estimator accounting for unequal sampling weights. Similarly, investigators will calculate the incidence rate of each CVD outcome among participants without the respective CVD at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNairy, MD, MSc, Principal Investigator — Washington University School of Medicine; Jean W Pape, MD, Principal Investigator — Weill Cornell Medical College /Les Centres GHESKIO
Locations (1):
- Les Centres GHESKIO, Port-au-Prince, West, Haiti

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data collected during the trial, after deidentification will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and SAP available after publication and ending 3 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal may have access. Proposals should be directed to the PI at mam9365@med.cornell.edu. To gain access, data requestors will need to sign a data access agreement. Data are available following publications through 3 years after publication and will be provided directly from the PI.

REFERENCES:
- [Background] Metz M, Pierre JL, Yan LD, Rouzier V, St-Preux S, Exantus S, Preval F, Roberts N, Tymejczyk O, Malebranche R, Deschamps MM, Pape JW, McNairy ML. Hypertension continuum of care: Blood pressure screening, diagnosis, treatment, and control in a population-based cohort in Haiti. J Clin Hypertens (Greenwich). 2022 Mar;24(3):246-254. doi: 10.1111/jch.14399. Epub 2022 Feb 24. PMID 35199944
- [Background] Sufra R, Lookens Pierre J, Dade E, Rouzier V, Apollon A, St Preux S, Preval F, Inddy J, Metz M, Tymejczyk O, Nash D, Malebranche R, Deschamps M, Pape JW, Goncalves MD, McNairy ML, Yan LD. Diabetes Epidemiology Among Adults in Port-au-Prince, Haiti: A Cross-Sectional Study. Front Endocrinol (Lausanne). 2022 Feb 24;13:841675. doi: 10.3389/fendo.2022.841675. eCollection 2022. PMID 35282460
- [Background] Clermont A, Sufra R, Pierre JL, Mourra MN, Fox EL, Rouzier V, Dade E, St-Preux S, Inddy J, Erline H, Obed FP, Yan LD, Metz M, Lee MH, Fitzgerald DW, Deschamps MM, Pape JW, McNairy ML. Dietary Risk Factors for Cardiovascular Disease among Low-Income Haitian Adults: Findings from a Population-Based Cohort. Nutrients. 2022 Feb 13;14(4):787. doi: 10.3390/nu14040787. PMID 35215437
- [Background] Yan LD, Rouzier V, Pierre JL, Lee MH, Muntner P, Parsons PJ, Apollon A, St-Preux S, Malebranche R, Pierre G, Emmanuel E, Nash D, Kingery J, Walsh KF, Smith CE, Metz M, Tymejczyk O, Deschamps M, Pape JW, Fitzgerald DW, McNairy ML. High Lead Exposure Associated With Higher Blood Pressure in Haiti: a Warning Sign for Low-Income Countries. Hypertension. 2022 Jan;79(1):283-290. doi: 10.1161/HYPERTENSIONAHA.121.18250. Epub 2021 Nov 17. PMID 34878898
- [Background] Lookens J, Tymejczyk O, Rouzier V, Smith C, Preval F, Joseph I, Baptiste RJ, Victor J, Severe P, Apollon S, Dumont E, Forestal G, St Preux S, Rivera V, Seo G, Charles B, Ariste W, Kingery J, Devieux J, Koenig S, Nash D, Fitzgerald D, Safford M, Deschamps MM, Pape J, McNairy M. The Haiti cardiovascular disease cohort: study protocol for a population-based longitudinal cohort. BMC Public Health. 2020 Nov 1;20(1):1633. doi: 10.1186/s12889-020-09734-x. PMID 33131500
- [Background] Yan LD, Lookens Pierre J, Rouzier V, Theard M, Apollon A, St Preux S, Kingery JR, Jamerson KA, Deschamps M, Pape JW, Safford MM, McNairy ML. Comparing six cardiovascular risk prediction models in Haiti: implications for identifying high-risk individuals for primary prevention. BMC Public Health. 2022 Mar 19;22(1):549. doi: 10.1186/s12889-022-12963-x. PMID 35305599
- [Background] Smith CE, Metz M, Lookens Pierre J, Rouzier V, Yan LD, Sufra R, Dade E, Preval F, Ariste W, Rivera V, Tymejczyk O, Peck R, Koenig S, Deschamps MM, Pape W, McNairy ML. Comparison of community and clinic-based blood pressure measurements: A cross-sectional study from Haiti. PLOS Glob Public Health. 2022;2(9):e0001064. doi: 10.1371/journal.pgph.0001064. Epub 2022 Sep 30. PMID 36285251
- [Background] Yan LD, Devieux JG, Pierre JL, Dade E, Sufra R, St Preux S, Tymejczyk O, Nash D, Metz M, Lee MH, Fitzgerald DW, Deschamps M, Pape JW, McNairy ML, Rouzier V. The relationship between perceived stress and support with blood pressure in urban Haiti: A cross-sectional analysis. PLOS Glob Public Health. 2022;2(5):e0000263. doi: 10.1371/journal.pgph.0000263. Epub 2022 May 2. PMID 35785017
- [Background] Dade E, Metz M, Pierre JL, Rouzier V, Sufra R, Fox E, Preval F, St-Preux S, Zephir JR 2nd, Ariste W, Rasul R, Sabwa S, Roberts N, Deschamps MM, Severe P, Fitzgerald D, Pape JW, Yan LD, McNairy ML. High prevalence of obesity among women in urban Haiti: Findings from a population-based cohort. Front Public Health. 2022 Oct 5;10:976909. doi: 10.3389/fpubh.2022.976909. eCollection 2022. PMID 36276356
- [Background] Clermont A, Rouzier V, Pierre JL, Sufra R, Dade E, Preval F, St-Preux S, Deschamps MM, Apollon A, Dupnik K, Metz M, Duffus Y, Sabwa S, Yan LD, Lee MH, Palmer LG, Gerber LM, Pecker MS, Mann SJ, Safford MM, Fitzgerald DW, Pape JW, McNairy ML. High Dietary Sodium, Measured Using Spot Urine Samples, is Associated with Higher Blood Pressure among Young Adults in Haiti. Glob Heart. 2023 Feb 14;18(1):5. doi: 10.5334/gh.1187. eCollection 2023. PMID 36817226
- [Background] Kingery JR, Roberts NL, Lookens Pierre J, Sufra R, Dade E, Rouzier V, Malebranche R, Theard M, Goyal P, Pirmohamed A, Yan LD, Hee Lee M, Nash D, Metz M, Peck RN, Safford MM, Fitzgerald D, Deschamps MM, Pape JW, McNairy M. Population-Based Epidemiology of Heart Failure in a Low-Income Country: The Haiti Cardiovascular Disease Cohort. Circ Cardiovasc Qual Outcomes. 2023 Feb;16(2):e009093. doi: 10.1161/CIRCOUTCOMES.122.009093. Epub 2022 Dec 6. PMID 36472189
- [Background] Rasul R, Rouzier V, Sufra R, Yan LD, Joseph I, Mourra N, Sabwa S, Deschamps MM, Fitzgerald DW, Pape JW, Nash D, McNairy ML. Extreme Food Insecurity and Malnutrition in Haiti: Findings from a Population-Based Cohort in Port-au-Prince, Haiti. Nutrients. 2022 Nov 17;14(22):4854. doi: 10.3390/nu14224854. PMID 36432540
- [Background] Yan LD, McNairy ML, Devieux JG, Pierre JL, Dade E, Sufra R, Gerber LM, Roberts N, St Preux S, Malebranche R, Metz M, Tymejczyk O, Nash D, Deschamps M, Safford MM, Pape JW, Rouzier V. Neighborhood cohesion and violence in Port-au-Prince, Haiti, and their relationship to stress, depression, and hypertension: Findings from the Haiti cardiovascular disease cohort study. PLOS Glob Public Health. 2022;2(7):e0000503. doi: 10.1371/journal.pgph.0000503. Epub 2022 Jul 27. PMID 36819610
- [Background] Yan LD, Sufra R, St Sauveur R, Jean-Pierre MC, Apollon A, Malebranche R, Theard M, Pierre G, Devieux J, Lau J, Mourra N, Roberts NLS, Rasul R, Nash D, Pirmohamed AM, Devereux RB, Lee MH, Kwan GF, Safford MM, Adrien L, Alfred JP, Deschamps M, Severe P, Fitzgerald DW, Pape JW, Rouzier V, McNairy ML; Haiti Cardiovascular Disease Cohort study team. Spectrum of prevalent cardiovascular diseases in urban Port-au-Prince, Haiti: a population-based cross-sectional study. Lancet Reg Health Am. 2024 Apr 4;33:100729. doi: 10.1016/j.lana.2024.100729. eCollection 2024 May. PMID 38590326
- [Background] Roberts NLS, Pierre JL, Rouzier V, Sufra R, St-Preux S, Yan LD, Metz M, Clermont A, Apollon A, Sabwa S, Deschamps MM, Kingery JR, Peck R, Fitzgerald D, Pape JW, Tummalapalli SL, McNairy ML. Prevalence and Severity of Chronic Kidney Disease in Haiti. Clin J Am Soc Nephrol. 2023 Jun 1;18(6):739-747. doi: 10.2215/CJN.0000000000000175. Epub 2023 Apr 18. PMID 37081617
- [Derived] Metz M, Sufra R, Ogyu A, Rouzier V, Sauveur RS, Celestin K, Forrestal G, Preval F, Jean M, Marcelin SE, Sarine A, Bennett C, Koenig S, Jamerson K, Pape JW, Yan LD, McNairy ML. Improvements in Blood Pressure Control and the Hypertension Care Continuum Over 2 Years in Urban Haiti Amidst Civil Unrest. J Clin Hypertens (Greenwich). 2025 Sep;27(9):e70153. doi: 10.1111/jch.70153. PMID 40991240
- [Derived] Rasul R, Sufra R, Pierre MCJ, St Sauveur R, Rouzier V, Inddy J, Hilaire E, Preval F, Yan LD, Mourra N, Ogyu A, Pierre DM, Pape JW, Nash D, McNairy ML. Prevalence of Cooking with Polluting Fuels and Association with Elevated Blood Pressure Among Adults in Port au Prince, Haiti: A Cross-Sectional Analysis. Glob Heart. 2025 Feb 28;20(1):22. doi: 10.5334/gh.1405. eCollection 2025. PMID 40026345
- [Derived] Sabwa S, Rouzier V, Sufra R, St Sauveur R, Mourra N, Rasul R, Inddy J, Yan LD, Sterling M, Pinheiro L, Deschamps M, Pape JW, McNairy ML. Cardiovascular Disease Multimorbidity and Decreased Health-Related Quality of Life in Haiti: A Cross-Sectional Study. J Am Heart Assoc. 2025 Feb 4;14(3):e036139. doi: 10.1161/JAHA.124.036139. Epub 2025 Jan 27. PMID 39868515
- [Derived] Yan LD, Rouzier V, Pierre JL, Dade E, Sufra R, Huffman MD, Apollon A, St Preux S, Metz M, Sabwa S, Morisset B, Deschamps M, Pape JW, McNairy ML. Polypill for atherosclerotic cardiovascular disease prevention in Haiti: Eligibility estimates in a low-income country. Front Epidemiol. 2022;2:925464. doi: 10.3389/fepid.2022.925464. Epub 2022 Jul 14. PMID 36816341